CLINICAL TRIAL: NCT03845569
Title: Impact of Habitual Protein Intake on Estimates of Dietary Protein Requirements in Resistance Trained Athletes
Brief Title: Influence of Habitual Protein Intake on AA Tracer Oxidation
Acronym: HPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Principle Investigator, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HPI
Record Dates: First submitted 2019-02-13; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Protein/Amino Acid Metabolism; Indicator Amino Acid Oxidation Method
Keywords: Amino acids; Protein; metabolism; IAAO; Tracer; Indicator amino acid; Resistance trained

STUDY DESIGN:
Intervention Model Description: Randomized crossover trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habitual Protein phase (Other): A trial investigating protein oxidation/metabolism that was used to model resistance trained individual's habitual dietary protein intake (2.2g/kg/d).
  Interventions: Other: Three day Controlled Diet
- Moderate Protein Phase (Experimental): A series of three trials over a one week period investigating protein oxidation/metabolism that was used to investigate the metabolic response of decreased protein intake (1.2g/kg/d) over a period of five days (trials on days 1, 3, 5 following reduction in protein intake from 2.2g/kg/d to 1.2g/kg/d) relative to the Habitual protein phase trial.
  Interventions: Other: Dietary protein intake reduction

INTERVENTIONS:
Other: Dietary protein intake reduction — Following two days of controlled diet at 2.2g/kg/d of dietary protein, intake was reduced to 1.2g/kg/d for five days, and protein metabolism was measured on days 1, 3, and 5.
  Arms: Moderate Protein Phase
Other: Three day Controlled Diet — Three days of a controlled diet providing 2.2g/kg/d of dietary protein with protein metabolism measured on day 3. This was used to model the habitual intake of this cohort.
  Arms: Habitual Protein phase

SUMMARY:
Protein is an essential nutrient that one's diet to maintain important bodily functions and to recover from exercise. Currently, the Indicator Amino Acid Oxidation method (IAAO) has been used to determine protein requirements in a variety of populations including children, neonates, the elderly and recently, resistance trained populations. This study serves to test the robustness of the IAAO method and to determine if high habitual dietary protein intake, as seen in resistance trained males, has the potential to influence the protein requirements determined by the IAAO method. Further, the current study also aims to determine how the body metabolizes or uses dietary protein and how it might change when consuming a protein intake that is less than what is habitually consumed.

DETAILED DESCRIPTION:
This study employed a two-phase randomized crossover design, where participants performed both a High/Habitual protein phase and a moderate protein phase. The Habitual protein phase is designed to model resistance trained individual's habitual protein consumption by providing 2.2g/kg/d in a controlled diet. The Moderate protein phase is designed to investigate the impact of decreasing dietary protein intake to a moderate amount (1.2g/kg/d) over five days on protein metabolism. Both phases used the stable isotope L-[1-13C]Phenylalanine and metabolic trails were modelled after the indicator amino acid oxidation (IAAO) technique.

High Protein Phase The high protein phase is three days in length, with diet-controlled throughout, and a metabolic trail on day 3. Participants will perform whole-body resistance exercise on days one and three.

Moderate protein phase The Moderate protein phase is seven days in length, with MT on days three, five and seven. Dietary intake will be controlled throughout the whole phase providing either 2.2 g/kg/d of protein (days one and two), or 1.2 g/kg/d (days three through seven). Full body resistance exercise will be performed performed on days one, three, five and seven.

This phase will allow measurement of protein metabolism over five days following a decrease in dietary protein intake, and to determine the effect of dietary changes on the IAAO method.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, weight-trained individuals that have trained consistently for > 1 year
* Habitually dietary protein consumption of 1.9 to 3.0g/kg/d
* Train each muscle group (i.e. chest, back, legs) at least twice a week
* Body mass stable in the last month
* Meets strength relative-to-weight guidelines (adapted from Morton et al., 2016; Chilibeck et -al., 1997)

  * Bench Press: - Bodyweight (kg) * 1.25
  * Leg Press: - Bodyweight (kg) *4.0

Exclusion Criteria:

* Inability to meet health and PA guidelines according to the PAR-Q+
* Inability to adhere to any of the protocol guidelines (e.g. alcohol and caffeine consumption)
* Regular tobacco use, screened by questionnaire
* Illicit drug use (e.g. growth hormone, testosterone, etc.), screened by a survey in training log

  * 1 month sedentary in the last 6 months prior to study participation
  * 30 minutes of continuous cardio per exercise session
* BMI > or equal to 35
* Individual plans to increase or decrease body mass in the next 3 months
* Use of supplements (excluding whey protein), such as creatine and beta-alanine, in the last 30 days

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Phenylalanine excretion (F13CO2) | Through study completion, an average of 3 months
  Expressed as µmol/kg/h; phenylalanine excretion is determined via breath enrichment (F13CO2) of the oral tracer. Breath 13CO2 enrichment was measured by continuous-flow isotope ratio mass spectrometry
Phenylalanine oxidation (PheOX) | Through study completion, an average of 3 months
  Expressed as µmol/kg/h; phenylalanine excretion is determined via breath and urine enrichment of the oral tracer. Breath 13CO2 enrichment was measured by continuous-flow isotope ratio mass spectrometry and urinary L-[1-13C] phenylalanine was measured by liquid chromatography tandem mass spectrometry

SECONDARY OUTCOMES:
Phenylalanine Rate of Appearance (PheRa/Flux) | Through study completion, an average of 3 months
  In µmol/kg/h; phenylalanine rate of appearance is determined via urinary enrichment of the oral tracer by liquid chromatography tandem mass spectrometry.
Net Protein Balance | Through study completion, an average of 3 months
  In µmol/kg/h; calculated as the difference between whole-body protein synthesis and protein breakdown. ). Breath 13CO2 enrichment was measured by continuous-flow isotope ratio mass spectrometry and urinary L-[1-13C] phenylalanine was measured by liquid chromatography tandem mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Moore, PhD, Principal Investigator — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Tinline-Goodfellow CT, West DWD, Malowany JM, Gillen JB, Moore DR. An Acute Reduction in Habitual Protein Intake Attenuates Post Exercise Anabolism and May Bias Oxidation-Derived Protein Requirements in Resistance Trained Men. Front Nutr. 2020 Apr 22;7:55. doi: 10.3389/fnut.2020.00055. eCollection 2020. PMID 32391374